CLINICAL TRIAL: NCT00022425
Title: Multiple-Dose Phase I and Pharmacokinetic Trial of Perillyl Alcohol
Brief Title: Perillyl Alcohol in Preventing Recurrent Breast Cancer in Women Who Have Been Treated With Surgery With or Without Adjuvant Therapy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Prevention
Other Study IDs: CDR0000068816; CCF-IRB-3574; CCF-N01-CN-55131; NCI-P01-0189
Record Dates: First submitted 2001-08-10; First posted 2003-01-27 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2003-09

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — perillyl alcohol

INTERVENTIONS:
Drug: perillyl alcohol

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the recurrence of cancer. The use of perillyl alcohol may be effective in preventing the recurrence of breast cancer.

PURPOSE: Phase I trial to study the effectiveness of perillyl alcohol in preventing the recurrence of breast cancer in women who have been treated with surgery with or without adjuvant therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of perillyl alcohol in women at risk for recurrent breast cancer.
* Determine the toxicity of this drug in these patients.
* Determine the single-dose and multiple-dose pharmacokinetics of this drug in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive oral perillyl alcohol once daily on days 1-28. Treatment continues every 4 weeks for 3 courses.

Cohorts of 6 patients receive escalating doses of perillyl alcohol until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience grade 1 toxicity or at least 1 of 6 patients experience grade 2 or greater toxicity.

Patients are followed weekly.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Personal history of stage Tis, I, II, or IIIA breast cancer
* Previously treated with definitive resection with curative intent
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* Over 18

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm3
* Platelet count at least 100,000/mm3
* Hemoglobin at least 9.0 g/dL

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* AST and ALT no greater than 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 1.5 times ULN

Renal:

* Creatinine no greater than 1.6 mg/dL

Other:

* No known malabsorption syndrome
* No contraindication to perillyl alcohol
* No hypersensitivity to citrus or soybean products
* No non-breast malignancy within the past 2 years except nonmelanoma skin cancer or carcinoma in situ
* No active malignancy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 6 months since prior chemotherapy

Endocrine therapy:

* Concurrent adjuvant hormonal therapy allowed

Radiotherapy:

* At least 6 months since prior radiotherapy

Surgery:

* See Disease Characteristics
* At least 6 months since prior surgery
* At least 2 years since prior primary surgery
* More than 4 weeks since prior surgery requiring general anesthesia, including breast reconstructive surgery

Other:

* More than 3 months since prior enrollment in a single-dose study of perillyl alcohol
* More than 3 months since prior enrollment in current study (at a lower dose level)
* No concurrent vitamin supplements except a daily multivitamin (recommended daily allowance)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-06

CONTACTS AND LOCATIONS:
Overall Officials: George Thomas Budd, MD, Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio, United States